CLINICAL TRIAL: NCT06193590
Title: Safety and Efficacy of a Suction Cervical Stabilizer Compared to the Standard Tenaculum for Intrauterine Procedures in the Clinic Setting
Brief Title: Suction Cervical Stabilizer Compared to Standard Tenaculum for Intrauterine Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Alissa M Conklin, Assistant Professor of Clinical Obstetrics and Gynecology, Indiana University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19699
Record Dates: First submitted 2023-12-04; First posted 2024-01-05 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Intrauterine Device (IUD); Abnormal Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Carevix (Experimental): suction cervical stabilizer utilized for intrauterine procedures
  Interventions: Device: Carevix
- Tenaculum (Active Comparator): standard of care cervical stabilization device
  Interventions: Device: Tenaculum

INTERVENTIONS:
Device: Carevix — Cervical stabilization device that uses vacuum
  Arms: Carevix
Device: Tenaculum — standard of care cervical stabilization device
  Arms: Tenaculum

SUMMARY:
To evaluate patient-reported pain, bleeding, and device efficiency along with provider satisfaction and ease of use between intrauterine procedures employing a suction cervical stabilizer (new device, FDA approved, atraumatic) or single-tooth tenaculum (standard, traumatic). This device, cleared by the FDA in 2023, was studied in Europe and showed pain reduced by up to 73% and bleeding reduced by 78% compared to the single-tooth tenaculum for intrauterine contraceptive device insertion. The investigators seek to study this device in the United States, and trial it among all intrauterine procedures.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 years or older

  * Speaks and reads in English
  * Able to consent on their own
  * Will undergo any intrauterine procedure using the Carevix (for exposure group) or using Tenaculum (for Control Group)
  * Cervix at least 26 mm in diameter
  * Twenty providers performing this procedure

Exclusion Criteria:

* • Vaginal bleeding of unknown origin

  * Cervix less than 26 mm in diameter
  * Nabothian cyst on anterior lip of cervix
  * Cervical myomas
  * Cervical abnormalities
  * Pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alissa Conklin, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yaron M, Legardeur H, Barcellini B, Akhoundova F, Mathevet P. Safety and efficacy of a suction cervical stabilizer for intrauterine contraceptive device insertion: Results from a randomized, controlled study. Contraception. 2023 Jul;123:110004. doi: 10.1016/j.contraception.2023.110004. Epub 2023 Mar 11. PMID 36914147
- See also: journal article — https://pubmed.ncbi.nlm.nih.gov/36914147/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from a women's health clinic in Indianapolis. Enrolled participants were at least 18 years old, English-speaking, and scheduled to undergo an intrauterine procedure. A total of 73 patients were enrolled with 60 eligible participants who received cervical stabilization during their procedure.
Pre-assignment Details: Patients were ineligible if they did not meet these criteria, as well as if they presented with vaginal bleeding of unknown origin, cervix less than 26 mm in diameter, Nabothian cyst on anterior lip of cervix, cervical myomas, cervical abnormalities/shape, or if they were pregnant. Patients were also designated ineligible if they did not receive any cervical stabilization. Patients were recruited in two waves corresponding with each arm.
Period: Overall Study
Arm/Group | Carevix | Tenaculum
Started | 36 | 37
Completed | 30 | 30
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carevix | Tenaculum | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Customized [Count of Participants; unit: Participants]
  Age (years): 18-19 | 0 | 1 | 1
  Age (years): 20-30 | 14 | 6 | 20
  Age (years): 31-40 | 8 | 11 | 19
  Age (years): 41-50 | 6 | 8 | 14
  Age (years): 51-60 | 1 | 2 | 3
  Age (years): 61+ | 1 | 1 | 2
  Age (years): Missing | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Marital Status [Count of Participants; unit: Participants]
  Single | 13 | 13 | 26
  Domestic partnership (or living together but not married) | 5 | 2 | 7
  Married | 10 | 13 | 23
  Divorced | 1 | 2 | 3
  Widowed | 1 | 0 | 1
  Other | 0 | 0 | 0
  Prefer not to say | 0 | 0 | 0
Highest level of complete education [Count of Participants; unit: Participants]
  Less than High School | 0 | 1 | 1
  High School, GE, or equivalent | 11 | 5 | 16
  Some college | 0 | 5 | 5
  Associate, Technical, or 2 year degree | 3 | 3 | 6
  Bachelor's or 4 year degree | 10 | 9 | 19
  Master's degree | 3 | 5 | 8
  Doctorate | 1 | 2 | 3
  License or Professional Certification | 0 | 0 | 0
  Other | 2 | 0 | 2
  Prefer not to say | 0 | 0 | 0
Employment Status [Count of Participants; unit: Participants]
  Unemployed | 3 | 3 | 6
  Student | 3 | 1 | 4
  Part-time (less than 40 hours a week) | 3 | 1 | 4
  Full-time (40+ hours a week) | 16 | 19 | 35
  Self-employed, Freelance, or Contractor | 2 | 3 | 5
  Retired | 1 | 1 | 2
  Other | 0 | 0 | 0
  Prefer not to say | 1 | 0 | 1
  Student and Part-time | 0 | 1 | 1
  Student and Full-time | 0 | 1 | 1
  Missing | 1 | 0 | 1
Nulliparous/Multiparous [Count of Participants; unit: Participants]
  Nulliparous | 12 | 13 | 25
  Multiparous | 18 | 17 | 35
  Vaginal delivery | 14 | 16 | 30
  Caesarean Section delivery | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Patient-perceived Pain
Description: Patients will be asked to rate their pain using the Numeric Rating Scale, a pain screening tool commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable". Participants fill out their survey once the procedure and clinical appointment is concluded.
Time Frame: Immediately after intrauterine procedure and scheduled appointment is complete (approx. 5-10 minutes after procedure completion)
Population: Participants who underwent an intrauterine procedure with either the Carevix device or the Tenaculum.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Carevix | Tenaculum
Number analyzed (Participants) | 30 | 30
score on a scale | 3 [2 to 4.75] | 4 [2 to 7]
Statistical Analysis 1: Comparison: Carevix vs Tenaculum; Test type: Superiority; p = 0.21, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Provider-perceived Bleeding
Description: Bleeding perceived by the provider during and after the procedure.
Time Frame: as for outcome 1
Population: Providers who completed the intrauterine procedure with their respective participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Carevix | Tenaculum
Number analyzed (Participants) | 30 | 30
Participants
  Had to manage/stop bleeding on cervical tissues | 3 | 9
  Did not have to manage/stop bleeding | 27 | 21
Statistical Analysis 1: Comparison: Carevix vs Tenaculum; Test type: Superiority; p = 0.1, Fisher Exact

3. Secondary Outcome: Provider-perceived Ease of Use
Description: Providers will report their perceived ease of use with the Carevix device indicating "Strongly Disagree, Disagree, Agree, or Strongly Agree" and open response.
Time Frame: as for outcome 1
Population: Providers were only asked about the "Ease of use" for the Carevix device.
Measure: Count of Participants; unit: Participants
Arm/Group | Carevix
Number analyzed (Participants) | 30
Participants
  Strongly Agree | 12
  Agree | 17
  Disagree | 1
  Strongly Disagree | 0
  I don't know/Not sure | 0

4. Secondary Outcome: Provider-perceived Satisfaction
Description: Providers will report their perceived satisfaction indicating "Strongly Disagree, Disagree, Agree, or Strongly Agree" and open response. In the Tenaculum arm, providers reported if they preferred the cervical tenaculum to the Carevix device. Providers complete their portion of the survey after the appointment is concluded.
Time Frame: as for outcome 1
Population: Providers who completed the intrauterine procedure with their respective participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Carevix | Tenaculum
Number analyzed (Participants) | 30 | 30
Participants
  Strongly Agree | 14 | 2
  Agree | 10 | 8
  I don't know not sure | 0 | 16
  Disagree | 5 | 3
  Strongly Disagree | 1 | 1
Statistical Analysis 1: Comparison: Carevix vs Tenaculum; Test type: Superiority; p = 0.001, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were assessed by providers during follow-up visits or patient reported, up to 2-months post-procedure.
Arm/Group | Carevix | Tenaculum
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/37
Other Adverse Events (participants affected / at risk) | 0/36 | 0/37

LIMITATIONS AND CAVEATS:
Not all clinic providers wanted to participate in the trial which hindered recruitment. Similarly, not all providers consistently utilized ANY cervical stabilization which rendered otherwise eligible participants unable to continue in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT06193590/Prot_SAP_000.pdf
  • Informed Consent Form: Carevix arm ICF (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT06193590/ICF_001.pdf
  • Informed Consent Form: Tenaculum arm ICF (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT06193590/ICF_002.pdf